CLINICAL TRIAL: NCT05965726
Title: RECOVER-VITAL: A Platform Protocol for Evaluation of Interventions for Viral Persistence, Viral Reactivation, and Immune Dysregulation in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-VITAL: Platform Protocol, Appendix to Measure the Effects of Paxlovid on Long COVID Symptoms
Acronym: RECOVER-VITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kanecia Obie Zimmerman (Other)
Responsible Party: Sponsor-Investigator, Kanecia Obie Zimmerman, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00111697_A; OTA-21-015G (Other Grant/Funding Number: NIH grant to RTI; RTI subcontracting with DCRI)
Record Dates: First submitted 2023-07-25; First posted 2023-07-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Long COVID-19; Long COVID
Keywords: PASC; Paxlovid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — nirmatrelvir and ritonavir drug combination; Ritonavir

STUDY DESIGN:
Intervention Model Description: As part of screening, potential participants will answer symptom questions. Eligible participants will then complete relevant Symptom Cluster assessments at the Screening visit. Participants will subsequently be assigned to one of the three Symptom Clusters based on the assessments.
  Participants must meet certain criteria within a specific symptom cluster in order to be included in the cluster. After study enrollment and initial cluster assignment, further assessments will be performed. Participants will undergo assessments for the symptom clusters for which the participants qualify.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Paxlovid 25 day dosing (Experimental): Paxlovid (nirmatrelvir 300mg, ritonavir 100mg) BID (twice a day) x 25 days
  Interventions: Drug: Paxlovid 25 day dosing
- Paxlovid 15 day dosing (Experimental): Paxlovid (nirmatrelvir 300mg, ritonavir 100mg) BID (twice a day) x 15 days then ritonavir 100mg plus nirmatrelvir-matching placebo x 10 days
  Interventions: Drug: Paxlovid 15 day dosing
- Ritonavir plus nirmatrelvir-matching placebo (Placebo Comparator): Ritonavir 100mg plus nirmatrelvir-matching placebo BID (twice a day) x 25 days
  Interventions: Drug: Ritonavir plus nirmatrelvir-matching placebo

INTERVENTIONS:
Drug: Paxlovid 25 day dosing — Nirmatrelvir 300mg and ritonavir 100mg taken BID (twice a day) for 30 days
  Arms: Paxlovid 25 day dosing
Drug: Paxlovid 15 day dosing — Nirmatrelvir 300mg and ritonavir 100mg taken BID (twice a day) for 15 days then ritonavir 100mg taken BID plus nirmatrelvir matching placebo BID for 15 days
  Arms: Paxlovid 15 day dosing
Drug: Ritonavir plus nirmatrelvir-matching placebo — Ritonavir 100mg taken BID (twice a day) plus nirmatrelvir matching placebo BID for 30 days
  Arms: Ritonavir plus nirmatrelvir-matching placebo

SUMMARY:
This is an appendix of master protocol (NCT05595369) designed to be flexible so that it is suitable for a wide range of settings within health care systems and in community settings where it can be integrated into COVID-19 programs and subsequent treatment plans. This sub-study is a prospective, multi-center, double-blind, randomized, controlled trial evaluating nirmatrelvir/ritonavir (Paxlovid) in two dosing durations for the treatment of Post-Acute Sequelae of SARS-CoV-2 Infection (PASC). The study is evaluating potential mechanisms of action, efficacy, and safety of antivirals and other therapeutics in individuals with PASC, according to the platform protocol objectives. The hypothesis is that persistent viral infection and/or overactive/chronic immune response and inflammation are underlying contributors to PASC and that antiviral and other applicable therapies may result in viral clearance or decreased inflammation and improvement in PASC symptoms.

DETAILED DESCRIPTION:
For this appendix of the master protocol (NCT05595369), participants will be randomized to Paxlovid (nirmatrelvir/ritonavir) vs. ritonavir control plus nirmatrelvir-matching placebo.

When there are multiple study interventions (sub-studies) available under the master protocol (NCT05595369), randomization will occur based on the specific inclusion/exclusion criteria of each appendix.

ELIGIBILITY:
See NCT NCT05595369 for RECOVER-VITAL: Platform Protocol level exclusion criteria which applies to this appendix

Additional Appendix Level Exclusion Criteria:

1. Known pregnancy*
2. Active or expected breastfeeding during the study
3. Known eGFR < 30 mL/min
4. Known severe hepatic impairment (Child-Pugh Class C)
5. Current use of drugs highly dependent on CYP3A for clearance** and for which elevated concentrations are associated with serious and/or life-threatening reactions and which cannot be interrupted during the time of study administration and within seven days before and after study drug administration
6. Current use of potent CYP3A inducers** where significantly reduced nirmatrelvir or ritonavir plasma concentrations may be associated with the potential for loss of virologic response and possible resistance

   * A pregnancy test must be performed at the Baseline Visit for participants who are capable of becoming pregnant.

     * A guide of drugs that may be contraindicated are listed in Section 4 CONTRAINDICATIONS of the Full Prescribing Information of the EUA for PAXLOVID. https://labeling.pfizer.com/ShowLabeling.aspx?id=16474&format=pdf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Change in cognitive dysfunction symptom cluster, as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) cognitive function T-score | Baseline to Day 90
  The PROMIS cognitive function-8a (PRO assessment) T-score is a quantitative measure of current cognitive function.
  The primary endpoint for cognitive dysfunction is improvement of at least 5 T-score points on the PROMIS-cognitive function as measured at 90 days compared to baseline.
Change in autonomic dysfunction symptom cluster, as measured by the orthostatic hypotension questionnaire (OHQ) | Baseline to Day 90
  The OHQ [Orthostatic Hypotension Questionnaire [PRO assessment)] is a measure of orthostatic intolerance, which has been the primary presentation of patients with PASC-related autonomic dysfunction. This measure includes the Orthostatic Intolerance Daily Activity Scale (OIDAS) and the Orthostatic Intolerance Symptom Assessment (OISA).
  The primary endpoint for autonomic dysfunction is improvement in autonomic function as defined by a ≥ 1-point decrease in the OHQ question 1 at 90 days compared to baseline.
Change in exercise intolerance symptom cluster, as measured by the Modified Depaul Symptom Questionnaire-Post Exertional Malaise (DSQ-PEM) | Baseline to Day 90
  DSQ-PEM assesses symptom frequency and severity over a 6-month look back period, however, for the purposes of this study, it will be modified to assess over a 1-week look back period. Frequency is rated on a 5-point Likert scale: 0 = none of the time, 1 = a little of the time, 2 = about half the time, 3 = most of the time, and 4 = all of the time. Severity is also rated on a 5-point Likert scale: 0 = symptom not present, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
  For exercise intolerance, the primary endpoint is improvement in PEM, defined as having no symptoms of moderate or greater severity with 50% or more frequency as determined by the DSQ-PEM short form at day 90.

SECONDARY OUTCOMES:
Change in cognitive dysfunction symptom cluster, as measured by a neurocognitive battery | Baseline to Day 90
  The neurocognitive battery outcome is a binary indicator of whether the participant has evidence of deficits (at least one standard deviation below the mean on at least one test within the battery).
Change in autonomic dysfunction symptom cluster, as measured by the active stand test | Baseline to Day 90
  The active stand test outcome is a binary indicator of whether the follow-up active stand test result was abnormal or normal.
Change in exercise intolerance symptom cluster, as measured by the endurance shuttle walk test (ESWT) | Baseline to Day 90
  The ESWT [endurance shuttle walk test (performance measure)] consists of timed walking on a 10m course.The ESWT will primarily be analyzed as a binary endpoint defined as an increase of at least 3 minutes of walking time at follow-up compared to baseline.
Occurrence of individual SAEs | Baseline to Day 190
Occurrence of one or more SAEs | Baseline to Day 190
Occurrence of AEs and SAEs leading to discontinuation | Baseline to Day 25
Occurrence of Events of Special Interest (ESIs) | Baseline to Day 190
Adherence in intervention versus control groups as measured by number of missed doses | Baseline to Day 25

CONTACTS AND LOCATIONS:
Locations (1):
- All sites listed under NCT05595369, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will share the summary of results on the study website: https:// recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT05965726/ICF_000.pdf